CLINICAL TRIAL: NCT02092441
Title: Inhalation Intervention for Nausea in the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michael D. April, Residency Associate Program Director for Research, Brooke Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: BAMC 395266-1
Record Dates: First submitted 2014-03-18; First posted 2014-03-20 (Estimated); Results first posted 2015-07-31 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-04

CONDITIONS: Nausea; Vomiting
Keywords: Nausea; Vomiting; Antiemetic
MeSH Terms: conditions — Nausea; Vomiting | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alcohol prep pad group (Active Comparator): isopropyl alcohol prep pad
  Interventions: Other: Alcohol prep pad group
- Normal Saline prep pad (Placebo Comparator): normal saline prep pad
  Interventions: Other: Normal Saline prep pad

INTERVENTIONS:
Other: Alcohol prep pad group — Subjects inhale scent of alcohol pad
  Arms: Alcohol prep pad group
Other: Normal Saline prep pad — Subjects inhale scent of placebo (normal saline) pads
  Arms: Normal Saline prep pad

SUMMARY:
Randomized controlled trial comparing inhalation of isopropyl alcohol vs placebo (normal saline) pads to treat nausea in emergency department patients.

DETAILED DESCRIPTION:
This study is to investigate if inhaling the scent of a typical medical alcohol prep pad will alleviate nausea as compared to a identically packaged normal saline prep pad for the Emergency Department patient with nausea. The study length will be 10 minutes long. The subjects will take several deep nasal inhalations at the 0, 2, 5 minute marks. Level of nausea will be recorded during these times and at 10 minutes. The investigators will also assess satisfaction of the intervention. As in previous post operative unit studies,the hypothesis is that there will a significant difference in levels of nausea between the alcohol pad group versus the normal saline pad group.

ELIGIBILITY:
Inclusion Criteria:

* age range of 18-65 years of age
* complaint of nausea and or vomiting
* ability to breathe through nose
* ability to read and write English

Exclusion Criteria:

* allergy to isopropyl alcohol
* pregnancy or pregnancy status unknown to subject. Pregnancy test only if part of clinical course.
* recent upper respiratory infection
* recent intake of cefoperazone, disulfiram, or metronidazole or any other medications that are known produce nausea when exposed to alcohol.
* use of antiemetic or psychoactive drug within 24 hours
* alcohol abuse
* nicotine within last 4 hrs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-04; Primary Completion 2014-11 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth L Beadle, MPAS, BS, Principal Investigator — BAMC; Curtis J Hunter, M.D., Study Director — BAMC
Locations (1):
- Emergency Department, Brooke Army Medical Center, Fort Sam Houston, Texas, United States

REFERENCES:
- [Background] Burleigh-Flayer HD, Gill MW, Strother DE, Masten LW, McKee RH, Tyler TR, Gardiner T. Isopropanol 13-week vapor inhalation study in rats and mice with neurotoxicity evaluation in rats. Fundam Appl Toxicol. 1994 Oct;23(3):421-8. doi: 10.1006/faat.1994.1123. PMID 7835543
- [Background] Gill MW, Burleigh-Flayer HD, Strother DE, Masten LW, McKee RH, Tyler TR, Gardiner TH. Isopropanol: acute vapor inhalation neurotoxicity study in rats. J Appl Toxicol. 1995 Mar-Apr;15(2):77-84. doi: 10.1002/jat.2550150204. PMID 7782562
- [Background] Burleigh-Flayer H, Garman R, Neptun D, Bevan C, Gardiner T, Kapp R, Tyler T, Wright G. Isopropanol vapor inhalation oncogenicity study in Fischer 344 rats and CD-1 mice. Fundam Appl Toxicol. 1997 Apr;36(2):95-111. doi: 10.1006/faat.1996.2284. PMID 9143479
- [Background] Cotton JW, Rowell LR, Hood RR, Pellegrini JE. A comparative analysis of isopropyl alcohol and ondansetron in the treatment of postoperative nausea and vomiting from the hospital setting to the home. AANA J. 2007 Feb;75(1):21-6. PMID 17304779
- [Background] Winston AW, Rinehart RS, Riley GP, Vacchiano CA, Pellegrini JE. Comparison of inhaled isopropyl alcohol and intravenous ondansetron for treatment of postoperative nausea. AANA J. 2003 Apr;71(2):127-32. PMID 12776641
- [Background] Pellegrini J, DeLoge J, Bennett J, Kelly J. Comparison of inhalation of isopropyl alcohol vs promethazine in the treatment of postoperative nausea and vomiting (PONV) in patients identified as at high risk for developing PONV. AANA J. 2009 Aug;77(4):293-9. PMID 19731848
- [Background] Wang SM, Hofstadter MB, Kain ZN. An alternative method to alleviate postoperative nausea and vomiting in children. J Clin Anesth. 1999 May;11(3):231-4. doi: 10.1016/s0952-8180(99)00035-5. PMID 10434220
- [Derived] Beadle KL, Helbling AR, Love SL, April MD, Hunter CJ. Isopropyl Alcohol Nasal Inhalation for Nausea in the Emergency Department: A Randomized Controlled Trial. Ann Emerg Med. 2016 Jul;68(1):1-9.e1. doi: 10.1016/j.annemergmed.2015.09.031. Epub 2015 Dec 8. PMID 26679977

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Alcohol Prep Pad Group | Normal Saline Prep Pad
Started | 37 | 43
Completed | 37 | 43
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alcohol Prep Pad Group | Normal Saline Prep Pad | Total
Number analyzed (Participants) | 37 | 43 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.65116 (14.17557) | 31.94595 (12.12652) | 33.9375 (13.3154)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 33 | 56
  Male | 14 | 10 | 24

OUTCOME MEASURES:

1. Primary Outcome: Nausea Verbal Numerical Rating Scale (0-10) at 10 Minutes Post Intervention
Description: Primary outcome is nausea and vomiting measured on a scale from 0 ("no nausea") to 10 ("worst nausea imaginable") Verbal Numerical Response Scale (VNRS) at 10 minutes post intervention.
Time Frame: 10 minutes post intervention
Measure: Median (Inter-Quartile Range); unit: VNRS
Arm/Group | Alcohol Prep Pad Group | Normal Saline Prep Pad
Number analyzed (Participants) | 37 | 43
VNRS | 3 [2 to 5] | 6 [4.5 to 8]

2. Secondary Outcome: Verbal Numerical Rating Scale Pain Score (0-10) at 10 Minutes Post Intervention
Description: Scale ranges from 0 ("no pain") to 10 ("worst pain imaginable")
Time Frame: 10 minutes post intervention
Measure: Median (Inter-Quartile Range); unit: VNRS
Arm/Group | Alcohol Prep Pad Group | Normal Saline Prep Pad
Number analyzed (Participants) | 37 | 43
VNRS | 6 [4 to 7] | 6 [2 to 7.5]

3. Other Pre Specified Outcome: Satisfaction Measured on a 5-point Likert Scale
Description: Patient satisfaction of smelling prep pad to alleviate nausea on a scale from 1 ("completely unsatisfied") to 5 ("completely satisfied")
Time Frame: 10 minutes post intervention
Measure: Median (Inter-Quartile Range); unit: 5 point Likert Scale
Arm/Group | Alcohol Prep Pad Group | Normal Saline Prep Pad
Number analyzed (Participants) | 37 | 43
5 point Likert Scale | 4 [3 to 5] | 2 [1 to 3]

ADVERSE EVENTS:
Arm/Group | Alcohol Prep Pad Group | Normal Saline Prep Pad
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/43
Other Adverse Events (participants affected / at risk) | 0/37 | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes